CLINICAL TRIAL: NCT05788445
Title: A Double-blind Randomized Controlled Clinical Trial of High-frequency nrTMS on the Contralateral Broca Mirror Area for Language Recovery in Patients With Non-fluent Aphasia After Glioma Surgery
Brief Title: High-frequency nrTMS on the Contralateral Broca Mirror Area for Glioma Patients With Early Postoperative Aphasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: No. 82203170
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Non-fluent Aphasia; Glioma
Keywords: human; language recovery; neuronavigated repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Aphasia, Broca; Glioma

STUDY DESIGN:
Intervention Model Description: There are two groups in this study. One group includes patients who receive nrTMS stimulation with high frequency on the contralateral Broca's area on the right hemisphere. The second group includes patients who receive nrTMS sham stimulation with high frequency on the contralateral Broca's area on the right hemishere.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There are two stimulating colis with the same shape, color and touch. The one is able to stimulate, the other is able to sham-stimulate. All patients are randomly assigned to use one of the two coils for treatment. Except for the designer, all participant, care provider, investigator, and outcomes assessorthey don not know who used which coil to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nrTMS treatment (Experimental): using nrTMS coli to stimulate the contralateral Broca's area on the right hemisphere with high freqency stimulation.
  Interventions: Device: nrTMS treatment
- nrTMS sham (Sham Comparator): using nrTMS sham-coli to stimulate the contralateral Broca's area on the right hemisphere with high frequency stimulation.
  Interventions: Device: nrTMS sham

INTERVENTIONS:
Device: nrTMS treatment — Using the nrTMS treatment coli to stimulation with high frequency
  Arms: nrTMS treatment
Device: nrTMS sham — Using the nrTMS sham coli to stimulation with high frequency
  Arms: nrTMS sham

SUMMARY:
The goal of this randomized clinical controlled trial is to determine whether the application of high frequency neuronavigated repetitive transcranial magnetic stimulation (nrTMS) on the contralateral of Broca's area can ameliorate glioma patients's non-fluent aphasia after tumor resection.

The questions this trial is aiming to answer are:

1. Whether the nrTMS can ameliorate glioma patients' postoperative language impairements.
2. if yes, how effective nrTMS is for improving glioma patients' postoperative language function.

DETAILED DESCRIPTION:
The including criteria:

A. Right-handed, age: 20~65 years old, tumor involves left language function area, no previous history of treatment of neurological diseases, and preoperative cognitive and language function assessment is normal B. Access to formal education at the primary level and above C. Postoperative pathology is primary low-grade glioma D. Language function assessed as motor aphasia on days 7-10 after surgery E. Willing to receive nrTMS rehabilitation F. The patient and family sign informed consent

The excluding criteria:

A. Tumor grows across the midline to the opposite side B. Undergoing unplanned surgery after the first tumor resection C. Patients request to withdraw from the study during treatment D. During the treatment period, the patient is unable to continue treatment due to force majeure E. Patient loss or refusal of follow-up during the study F. Patients are considered by the investigator to be unsuitable for participation in this study

All patients will receive nrTMS treatment or nrTMS sham treatment for 7 sessions within 10 days (one session per day), start at the 7th - 10th day after glioma resection. The effects of nrTMS treatment will be determine by using the Western Aphasia Battery to evaluate patients' language function after each session and each follow-up interview (every 7-10 days after the whole treatment session finished until the end of the 3rd month after tumor resection or patients' language evaluation shows the language function recoveried to the normal level).

ELIGIBILITY:
Inclusion Criteria:

A. Right-handed, age: 20~65 years old, tumor involves left language function area, no previous history of treatment of neurological diseases, and preoperative cognitive and language function assessment is normal B. Access to formal education at the primary level and above C. Postoperative pathology is primary low-grade glioma D. Language function assessed as motor aphasia on days 7-10 after surgery E. Willing to receive nrTMS rehabilitation F. The patient and family sign informed consent

Exclusion Criteria:

A. Tumor grows across the midline to the opposite side B. Undergoing unplanned surgery after the first tumor resection C. Patients request to withdraw from the study during treatment D. During the treatment period, the patient is unable to continue treatment due to force majeure E. Patient loss or refusal of follow-up during the study F. Patients are considered by the investigator to be unsuitable for participation in this study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Improvement of language function | from the day of tumor resection to 3 months after tumor resection
  Based on the result of western aphasia battery, patients' language score incrased 200% of the score before the treatment started.

SECONDARY OUTCOMES:
language recvoery | from the day of tumor resection to 3 months after tumor resection
  Based on the result of western aphasia battery, patients' language score increased above the cut off line for aphaisa that the language function can be identified as non-aphasia.